CLINICAL TRIAL: NCT00699621
Title: Platelet Transfusion in Acute Primary Intracerebral Hemorrhage for Patients on Platelet Inhibitors
Brief Title: Platelet Transfusion in Acute Intracerebral Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Oulu University Hospital (Matti Hillbom), Oulu University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-1 EUDRACT 2007-006206-24
Record Dates: First submitted 2008-06-12; First posted 2008-06-18 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral hemorrhage; Hematoma enlargement; Antiplatelet agent; Platelet transfusion; Outcome
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Platelet Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Platelet transfusion
  Interventions: Biological: platelets
- 2 (No Intervention): No platelet transfusion

INTERVENTIONS:
Biological: platelets — Four units of fresh platelets will be infused immediately
  Arms: 1

SUMMARY:
* To prove whether use of antiplatelet agents results into a rapid enlargement of hematoma after onset of acute intracerebral hemorrhage.
* To prove the efficacy and safety of platelet transfusion for prevention of hematoma growth in patients who were stricken by acute intracerebral hemorrhage while being on antiplatelet medication.

DETAILED DESCRIPTION:
* Hematoma growth is a well-known powerful determinant of mortality and poor outcome after intracerebral hemorrhage.
* Some observations suggest that previous use of antiplatelet agents associates with rapid hematoma enlargement and poor outcome after cerebral hemorrhage.
* Immediate platelet transfusion for such patients may prevent hematoma growth but also cause thromboembolic complications.

ELIGIBILITY:
Inclusion Criteria:

* being on either aspirin or clopidogrel or a combination of aspirin and dipyridamole
* acute primary ICH
* > 17 years
* admitted within 6 h after onset of ICH
* ICH score < 4

Exclusion Criteria:

* other type of ICH than acute primary intracerebral hemorrhage
* patients who need neurosurgery
* life expectancy less than 3 months due to comorbid disorders
* confirmed malignant disease (cancer)
* confirmed acute myocardial infarction
* hepatitis and/liver cirrhosis
* renal failure
* infectious disease (HIV, endocarditis etc.)
* current or previous hematologic disease
* women of childbearing age if pregnant
* participation in another study within the preceding 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Hematoma growth within 24 h measured as increase in hematoma volume observed by head CT | 24 hours

SECONDARY OUTCOMES:
Glasgow Outcome Score | 90 days
Cardiovascular death occurring within the treatment period | 90 days
Death due to any cause occurring within the treatment period | 90 days
Acute myocardial infarction | 90 days
Venous thromboembolism | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Matti E Hillbom, MD, PhD, Study Chair — Oulu University Central Hospital, Department of Neurology; Seppo S Juvela, MD, PhD, Study Director — Turku University Central Hospital, Department of Neurosurgery; Lauri Soinne, MD, PhD, Principal Investigator — Helsinki University Central Hospital, Department of Neurology; Olli Häppölä, MD, PhD, Study Director — Helsinki University Central Hospital; Aimo Rissanen, MD, PhD, Principal Investigator — Keski-Suomen Keskussairaala
Locations (1):
- Department of Neurology, Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112